CLINICAL TRIAL: NCT00751413
Title: A Multicenter, Open-Label, Single Dose Study to Evaluate the Safety, Tolerability and Plasma Concentration Profiles of MK0633 in Asthmatic Children Aged 6 to Less Than 12 Years
Brief Title: Plasma Levels of MK0633 in Children Ages 6-12 (0633-023)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0633-023; MK0633-023; 2008_529
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (1):
- 1 (Experimental): MK0633
  Interventions: Drug: Comparator: MK0633

INTERVENTIONS:
Drug: Comparator: MK0633 — A single dose of MK0633 10 mg or 25 mg film coated tablet. Dose will be based on patient weight.

SUMMARY:
To evaluate the safety, tolerability and plasma levels of single oral doses of MK0633 in pediatric asthma patients ages 6 to less than 12 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient has mild to moderate asthma
* Patient is able to swallow pills
* Patient is able to have have blood draws

Exclusion Criteria:

* Patient has required a visit to the hospital or emergency room due to an asthmatic event in the last 3 months
* Patient has an upper respiratory tract infection (URI)
* Patient has a history of stroke
* Patient consumes more than 4 caffeinated beverages per day

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single oral doses of MK0633 in pediatric asthma patients. | Physical examinations, vital sign measurements, laboratory safety tests (blood chemistry, hematology and urinalysis), urine ß-hCG test, and 12-lead ECGs will be performed at various scheduled time points throughout the study.

SECONDARY OUTCOMES:
To obtain information on plasma pharmacokinetics (e.g., AUC0-inf, Cmax, Tmax, apparent t½,) of MK0633 after a single oral dose administration in pediatric asthma patients | Plasma will be analyzed at specific time-points for MK0633 concentrations. Urine will be collected for the measurement of LTE4 concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC